CLINICAL TRIAL: NCT06827912
Title: Comparison of Postoperative Analgesic Effects of Interscalene and Shoulder Anterior Capsule Block in Arthroscopic Rotator Cuff Operations
Brief Title: Comparison of Interscalene and Anterior Shoulder Capsule Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Bülent Meriç Çam, Specialist Doctor, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-106
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Pain Intensity Assessment; Interscalene Nerve Block; Shoulder Anterior Capsule Block (SHAC Block); Pericapsular Nerve Group Block (PENG)
Keywords: Pain Management; Interscalene Block; Shoulder Anterior Capsular Block; Pericapsuler nerve group block; SHAC; PENG; Rotator cuff repair
MeSH Terms: conditions — Agnosia | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interscalene Block Group (Active Comparator)
  Interventions: Procedure: Shoulder Anterior Capsule Block
- SHAC Block Group (Active Comparator)
  Interventions: Procedure: Interscalene Nerve Block

INTERVENTIONS:
Procedure: Interscalene Nerve Block — After sterile conditions are provided with the patient in the supine position, the brachial plexus will be identified in the supraclavicular fossa above the clavicle with ultrasonography. The transducer will be directed cephalad and 20 cc 0.5% bupivacaine will be applied to the interscalene space with a 50 mm block needle from the point where the C 5-6-7 nerve roots give the impression of a rosary bead between the anterior and medial scalene muscles.
  Arms: SHAC Block Group
Procedure: Shoulder Anterior Capsule Block — In pericapsular nerve block application, the patient will be placed in a supine position and the arm will be externally rotated and abducted to 45 degrees. After sterile conditions are provided, the humerus head, the tendon of the subscapularis muscle and the deltoid muscle above it will be identified with ultrasonography. 15 cc of 0.5% bupivacaine will be injected into the interfascial space between the deltoid muscle and the subscapularis muscle with a 22gauge 50 mm block needle. Then, the block needle will be directed deep into the subscapularis muscle and another 5 cc of 0.5% bupivacaine will be injected under the subscapularis muscle.
  Arms: Interscalene Block Group

SUMMARY:
Due to the development and easy availability of ultrasonography devices, regional nerve blocks are routinely used by anesthesiologists among multimodal analgesia techniques. Interscalene and supraclavicular nerve blocks are the leading regional anesthesia techniques for shoulder surgeries. However, due to the phrenic nerve involvement and loss of motor function in the upper extremity in these block techniques, new nerve blocks have been developed and used for postoperative analgesia. One of the blocks that has been used increasingly in shoulder region surgeries and does not cause phrenic nerve involvement is the shoulder anterior capsule block (SHAC). The aim of this study is to compare the postoperative analgesic effects of interscalene nerve block and SHAC block in patients undergoing arthroscopic rotator cuff repair surgery.

DETAILED DESCRIPTION:
Shoulder arthroscopy is one of the most frequently performed orthopedic procedures today. Although it is a minimally invasive procedure, it has been associated with severe postoperative shoulder pain and many techniques have been investigated for pain management. Today, anesthesiologists try to control postoperative pain well as one of the important components of enhanced recovery after surgery (ERAS), as this increases patient comfort and accelerates recovery. At the same time, opioids are tried to be avoided as much as possible while controlling pain due to their serious side effects. For these reasons, interscalene nerve block is frequently used in shoulder arthroscopy patients and provides highly effective and long-lasting postoperative analgesia. Interscalene block can also be used alone for surgical anesthesia in patients undergoing shoulder arthroscopic surgery and is accepted as the gold standard regional anesthesia technique. However, due to phrenic nerve involvement in interscalene block and loss of motor function in the upper extremity, new nerve blocks continue to be discovered for postoperative analgesia.

In 2020, Altinpulluk et al. showed that methylene blue applied to the deep subscapular muscle in a cadaver, between the humerus head and the area, stained the entire shoulder joint capsule and a certain amount of the axillary region, and they named this new block as pericapsular nerve block (PENG). Kupeli et al. and Ramudarai et al. applied the local anesthetic drug to the interfascial area between the deltoid muscle and the subscapular muscle and named this block as PENG block. The investigators think that this is the axillary nerve block with the Fajardo approach defined by Altınpulluk et al. Because in the cadaver study conducted by Gonzalez et al., it was shown that methylene blue applied between the deltoid muscle and the subscapular muscle did not spread to the pericapsular area. Nevertheless, postoperative analgesia was provided with the local anesthetic drug applied with both approaches and a motor protective effect was demonstrated. The injection made in both areas together can be called shoulder anterior capsule block (SHAC).

In our clinic, in our routine practice, the investigators perform the anesthesia procedure of patients who will undergo arthroscopic rotator cuff repair without general anesthesia, only with interscalene block. Since the SHAC block, which is a relatively new block mentioned above, does not provide sufficient surgical anesthesia on its own, patients must also be placed under general anesthesia. Our study aims to compare patients who have arthroscopic rotator cuff repair under general anesthesia with SHAC block and patients who have arthroscopic rotator cuff repair with interscalene block alone in terms of postoperative analgesia and motor-protective effects.

Materials and methods Ethics This double-blind, single-center, parallel-arm, randomized controlled study was approved by Hitit University Research Ethics Committee, numbered 2024-106. The study will be conducted at Amasya University Sabuncuoğlu Şerefeddin Education and Research Hospital.

Randomization and blinding Patients will be randomly assigned to two equal groups (ISC group or SHAC group) using a computer-assisted randomization method using the "Research Randomizer" program (www.randomizer.org), 46 patients in a 1:1 ratio. Due to the nature of the interventions, blinding will not be possible for the anesthesiologist administering the anesthesia. However, in order to minimize bias, the investigators responsible for the evaluation of postoperative recovery times, pain scores, and opioid-related side effects will be blinded to group assignment throughout the study.

Protocol All patients were subjected to standard monitoring procedures (ECG, pulse-oximetry, blood pressure measurement) as in routine anesthesia practices. Regional block application will be performed in both groups in the preoperative period. In the SHAC group, patients will be placed under general anesthesia after the block, while in the interscalene block group, surgery will be performed only with regional block. After the preoperative block application, patients will be taken to the operation room. An intravenous patient-controlled analgesia device will be attached during transfer to the ward and the patient will be instructed on how to use it. Anesthesia in the operation room will be performed with an intravenous injection of 0.02mg/kg midazolam, 1mcq/kg fentanyl, 2-3mg/kg propofol and 0.6mg/kg rocuronium for patients in the SHAC group. Following intubation, anesthesia will be maintained with the inhalation agent sevoflurane. The target Minimum Alveolar Concentration (MAC) value will be adjusted to 1 MAC. After the surgery is completed, inhalation agents will be stopped, patients will be administered 2-4 mg/kg sugammadex intravenously, which eliminates neuromuscular blockade, and extubated when sufficient tidal volume is spontaneously created. After sufficient anesthetic recovery, the patient will be taken to the recovery room, and when the Aldrete score reaches 10, the patient will be transferred to the ward. During transfer to the ward, an intravenous patient-controlled analgesia device will be attached and the patient will be instructed on how to use it.

Patient controlled analgesia drug dose and device settings: Fentanyl will be set to 5mcq/ml, without loading and continuous infusion dose, full dose will be set to 10mcq. Lockout time will be set to 20 minutes, 4hour limit will be set to 100mcq.

Sample Size Calculation:

Since there is no randomized study in the literature that will refer to the primary outcome of our study, Cohen's effect sizes were used as the effect size. Using an independent sample t-test in two groups, the sample size for both groups was 21, with an effect size of 0.8, a margin of error of 0.05, and a power of 0.80, and a total of 42 patients. When the drop out was taken as 10%, the sample size required for the study was found to be 46 patients. G*Power version 3.1.9.4 was used to calculate the sample size.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 patients who will undergo arthroscopic rotator cuff repair,
* Patients between the ages of 18-75

Exclusion Criteria:

* Allergy to local anesthetics
* Infection at the block site
* Neuropathy in the involved extremity
* History of chronic opioid use
* Revision surgery
* History of hepatic and renal failure
* History of peripheral neuropathy
* History of diabetes mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Postoperative 12th hour pain score | Postoperative 12th hour
  Postoperative 12th hour pain score (will be evaluated with Numeric Rating Scale) Higher scores indicate worse condition

SECONDARY OUTCOMES:
Postoperative 1, 2, 4, 8, 12, 16, 24, 48 hours pain score | Postoperative 1, 2, 4, 8, 12, 16, 24, 48 hours
  Postoperative 1, 2, 4, 8, 12, 16, 24, 48 hours pain score (to be evaluated with Numeric Rating Scale) Higher scores indicate worse condition
Amount of opioid consumption | in the first 24 hours postoperatively
  Amount of opioid consumption in the first 24 hours postoperatively
Complications related to opioid use | in the first 24 hours postoperatively
  Complications related to opioid use such as nausea, vomiting, itching
Elephant flexion motor strength evaluation | in the first 24 hours postoperatively
  Elephant flexion motor strength evaluation (1-5 points)
Surgeon satisfaction level with Likert scale | during surgery
  It will be done to show how satisfied the surgeon is with the anesthesia technique during the time period between the beginning and end of the operation. It will be evaluated between 0-5 points. Higher scores indicate higher satisfaction.
Patient satisfaction level with Likert scale | postoperative 24th hour
  It will be done to measure the patient's satisfaction with the surgery according to the level of pain in the 24-hour postoperative period. It will be evaluated between 0-5 points. Higher scores indicate higher satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital, Amasya, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamak Altinpulluk E, Teles AS, Galluccio F, Simon DG, Olea MS, Salazar C, Fajardo Perez M. Pericapsular nerve group block for postoperative shoulder pain: A cadaveric radiological evaluation. J Clin Anesth. 2020 Dec;67:110058. doi: 10.1016/j.jclinane.2020.110058. Epub 2020 Sep 26. No abstract available. PMID 32987232
- [Background] Kupeli I, Yazici Kara M. Anesthesia or analgesia? New block for shoulder surgery: pericapsular nerve group block. Braz J Anesthesiol. 2022 Sep-Oct;72(5):669-672. doi: 10.1016/j.bjane.2021.05.009. Epub 2021 Jun 9. PMID 34118263
- [Background] Galluccio F, Fajardo Perez M, Yamak Altinpulluk E, Hou JD, Lin JA. Evaluation of Interfascial Plane and Pericapsular Nerve Blocks to the Shoulder Joint: A Preliminary Analysis of Shoulder Anterior Capsular Block. Pain Ther. 2021 Dec;10(2):1741-1754. doi: 10.1007/s40122-021-00326-0. Epub 2021 Oct 20. PMID 34669181
- [Derived] Cam BM, Tuzen AS, Duran HT, Akdogan MA. Comparison of interscalene block versus shoulder anterior capsule block for postoperative pain management in rotator cuff surgery: a randomized controlled trial. BMC Anesthesiol. 2025 Sep 29;25(1):459. doi: 10.1186/s12871-025-03351-0. PMID 41023793